CLINICAL TRIAL: NCT04967001
Title: Efficacy of 68Ga PSMA PET in the Diagnosis of Lymph Node Metastasis in Patients With Prostate Cancer: a Single Center Prospective Randomized Controlled Trial
Brief Title: 68Ga-PSMA PET in the Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Qin Weijun, Professor and Director, Department of Urology, Xijing Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20212032-F-1
Record Dates: First submitted 2021-07-11; First posted 2021-07-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasms; Metastases; PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSMAPET-MRI (Experimental)
  Interventions: Diagnostic Test: PSMA PET
- MRI-PSMAPET (Experimental)
  Interventions: Diagnostic Test: PSMA PET

INTERVENTIONS:
Diagnostic Test: PSMA PET — 68Ga-PSMA PET

SUMMARY:
Efficacy of 68Ga PSMA PET / CT in the diagnosis of lymph node metastasis in patients with prostate cancer: a single center prospective randomized controlled trial.

To identify and compare the diagnostic efficacy of 68Ga-PSMA PET/CT and mpMRI for lymph nodes in patients with newly diagnosed prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* High risk localized/locally advanced prostate cancer patients who are candidates for radical prostatectomy plus bilateral extended PLND
* ISUP Gleason grade group ≥ 4

Exclusion Criteria:

* Prior history of any other cancer in the last 5 years excluding basal cell carcinoma Proven metastases in bones or other distant metastases
* General contra-indications for MRI (pacemaker, aneurysm clips, any form of metal in the body, severe claustrophobia)
* Serious concomitant systemic disorders that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study objectives
* Metal implants in the pelvic region which will deteriorate PET/MR/CT image quality.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of PSMA PET and combined PSMA PET/MRI or PSMA PET/CT | 2 years
  To compare the diagnostic accuracy of PSMA PET and combined PSMA PET/MRI or PET/CT to that of the current standard multiparametric MRI, using histopathology as the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No